CLINICAL TRIAL: NCT02183532
Title: Pharmacokinetics of Single and Multiple Oral Doses of 5 mg BI 1356 in Healthy Chinese Volunteers
Brief Title: Pharmacokinetics of Single and Multiple Oral Doses of BI 1356 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218.58
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (1):
- BI 1356 BS (Experimental)
  Interventions: Drug: BI 1356 BS

INTERVENTIONS:
Drug: BI 1356 BS — single dose
Drug: BI 1356 BS — multiple doses

SUMMARY:
Study to investigate the pharmacokinetics of BI 1356 after single and multiple oral doses of 5 mg in Chinese healthy subjects

ELIGIBILITY:
Inclusion Criteria:

Male and female Chinese healthy volunteers who meet the criteria below:

* Persons without clinically remarkable findings or clinically evident complications based on their concurrent illness, past medical history, physical examination, vital signs (blood pressure, pulse rate, and body temperature), 12-lead Electrocardiogram (ECG), and laboratory test results
* Age ≥18 and Age ≤45 years
* Body weight ≥50 kg with BMI ≥19 and BMI ≤24 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Persons who deviate from the norm, and who show clinical findings (Blood pressure (BP), Heart rate (HR), and ECG) on consultation
* Persons with any clinically significant complications
* Persons with gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immune, or hormonal disorders
* Persons with central nervous system disorders (e.g., epilepsy), mental disorders, or neurological disorders
* Persons with a history of significant orthostatic hypotension, syncopal attacks, or blackouts
* Persons with chronic infection or severe acute infection
* Persons with a history of severe allergy/hypersensitivity (including allergies to drugs or inactive ingredients)
* Persons who will have received a drug with a long half-life (more than 24 hours) within the month before treatment in this study, within a period 10 times longer than the half-life of each drug, or during the study
* Persons who will have received a drug that may theoretically affect the study results based on the information obtained at the time of preparation of the protocol, within the 10 days before treatment or during the study (e.g inhibitors or inducers of Pgp or CYP 3A4)
* Persons who will have participated in another trial of an investigational drug within the 4 months before treatment or during the study
* Smokers (who smoke more than 10 cigarettes, or 3 cigars, or 3 pipes per day)
* Persons who cannot abstain from smoking throughout the study
* Persons who undoubtedly abuse alcohol
* Persons who abuse drugs
* Persons who donate blood of 100 mL or more within the 4 weeks before treatment
* Persons who perform rigorous exercise (within the week before treatment or during the study)
* Persons with any laboratory test result outside the reference range and for whom the result is considered a clinically significant change
* Persons who cannot obey the dieting rules of the study centre
* Persons with any ECG value outside the reference range and who are of clinical importance. Examples include, but are not limited to, QRS interval >120 ms.
* Pre-menopausal women (last menstruation <1 year prior to the date of informed consent) who:

  * are nursing or pregnant
  * or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to periodic pregnancy testing during their participation in the trial. Acceptable methods of birth control include transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner. No exception will be made.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cmax,ss (Maximum measured concentration of the analyte in plasma at steady state) | up to day 19
AUCτ (Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 19

SECONDARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) at different time points after single and multiple doses | up to day 19
tmax (Time from dosing to maximum measured concentration) at different time points after single and multiple doses | up to day 19
AUC0-infinity (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single dose administration) | up to day 7
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of last quantifiable analyte plasma concentration after single dose administration) | up to day 7
AUC0-24 (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours after single dose administration) | up to 24 h after single dose administration
AUC0-72 (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 hours after single dose administration) | up to 72 h after single dose administration
λz (Terminal rate constant in plasma) at different time points after single and multiple doses | up to day 19
t1/2 (Terminal half-life of the analyte in plasma) at different time points after single and multiple doses | up to day 19
MRTpo (Mean residence time of the analyte in the body) at different time points after single and multiple doses | up to day 19
CL/F (Apparent clearance of the analyte in plasma after extravascular administration) at different time points after single and multiple doses | up to day 19
Vz/F (Apparent volume of distribution during the terminal phase λz following extravascular administration) at different time points after single and multiple doses | up to day 19
Aet1-t2 (Amount of analyte that is eliminated in urine from time point t1 to time point t2) at different time points after single and multiple doses | up to 168 h after first dose and up to 24 h after last dose
fet1-t2 (Fraction of analyte eliminated in urine from time point t1 to time point t2) at different time points after single and multiple doses | up to 168 h after first dose and up to 24 h after last dose
Cmin,ss (Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) for multiple doses | up to 144 h after last dose
Cavg,ss (Average concentration of the analyte in plasma at steady state) | up to 144 h after last dose
AUCτ,ss (Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 144 h after last dose
CLRt1-t2,ss (Renal clearance of the analyte at steady state from time point t1 to time point t2) | up to 144 h after last dose
Cpre (Predose concentration of the analyte in plasma) at different time points | up to 120 h after first of multiple doses
PTF (Peak-Trough Fluctuation) | up to 120 h after first of multiple doses
RA,Cmax (Accumulation ratio of the analyte in plasma after multiple dose administration over a uniform dosing interval τ) based on Cmax | up to day 19
RA,AUC (Accumulation ratio of the analyte in plasma after multiple dose administration over a uniform dosing interval τ) based on AUCτ | up to day 19
Number of patients with adverse events | up to 28 days
Number of patients with abnormal findings in physical examination | up to 25 days
Number of patients with abnormal changes in laboratory parameters | up to 25 days
Number of patients with clinically significant changes in Vital signs (blood pressure [BP], pulse rate [PR]) | up to 25 days
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 25 days